CLINICAL TRIAL: NCT02270814
Title: Phase 2 Single Arm Trial of Cisplatin, Nab-Paclitaxel, and Cetuximab (CACTUX) in Patients With Incurable Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Cisplatin, Nab-Paclitaxel, and Cetuximab (CACTUX) in Patients With Incurable Head and Neck Squamous Cell Carcinoma
Acronym: CACTUX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201410073
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Cisplatin; Carboplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CACTUX: nab-paclitaxel, cisplatin (or carboplatin), cetuximab (Experimental): Up to 6 cycles of CACTUX may be given. The CACTUX regimen consists of:
  * nab-paclitaxel given intravenously over 30 minutes on an outpatient basis on Days 1, 8, and 15 of each 21-day cycle followed by
  * cisplatin given intravenously over 60 minutes on an outpatient basis OR carboplatin AUC5 given intravenously over 30 minutes on an outpatient basis on Day 1 of each 21-day cycle followed by
  * cetuximab given intravenously on an outpatient basis of Days 1, 8, and 15 of each 21-day cycle
  * Cisplatin or carboplatin may be given at the discretion of the investigator.
  After the completion of 6 cycles of CACTUX, maintenance therapy will be given and consists of:
  * nab-paclitaxel given intravenously over 30 minutes on an outpatient basis on Days 1 and 8 of each 21-day cycle
  * cetuximab given intravenously on an outpatient basis on Days 1, 8, and 15 of each 21-day cycle
  Interventions: Drug: nab-paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Biological: Cetuximab

INTERVENTIONS:
Drug: nab-paclitaxel
  Other Names: Abraxane; Albumin-bound paclitaxel; Paclitaxel protein-bound
Drug: Cisplatin
  Other Names: Cisplatinum; CDDP; cis-DDP; cis-Diamminedichloroplatinum; cis-Platinum II; DDP
Drug: Carboplatin
  Other Names: Paraplatin®; CBDCA
Biological: Cetuximab
  Other Names: Erbitux®

SUMMARY:
The purpose of this research study is to look at the effect of a treatment regimen called CACTUX on head and neck cancer. The CACTUX regimen is a combination of three drugs called cisplatin, nab-paclitaxel, and cetuximab (although carboplatin may be given in place of cisplatin if participants have previously had problems receiving cisplatin). The use of nab-paclitaxel in this combination is different from routine care, in which a drug called 5FU is often given instead, but the investigators group has conducted previous research where the investigators incorporated nab-paclitaxel into routine treatment with cisplatin, 5FU, and cetuximab. The investigators are looking at the incidence of side effects with the CACTUX regimen as well as response of the disease and health status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed incurable HNSCC of the oral cavity, oropharynx, larynx, hypopharynx, and/or Level 1-3 neck node with non-skin SCC and unknown primary. "Incurable" is defined as metastatic disease or a local or regional recurrence in a previously irradiated site that is unresectable (or patient declines resection).
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam per RECIST 1.1.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Adequate hematologic, renal, and hepatic function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 mg/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN, alkaline phosphatase ≤ 2.5 x IULN, unless bone metastasis is present in the absence of liver metastasis
  * Creatinine at or below IULN (males 0.7-1.30 mg/dl; females 0.6-1.10 mg/dl) OR Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* At least 4 months since completion of curative therapy, if given previously.
* Availability of diagnostic tumor tissue specimens for correlative studies.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 3 months after completing treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior systemic therapy for incurable disease.
* Grade 2 or higher peripheral neuropathy at screening.
* A history of other malignancy ≤ 2 years previous; exceptions are malignancies with a negligible risk of metastasis or death (e.g., expected 5-year OS > 90%) that were treated with an expected curative outcome, such as squamous cell carcinoma of the skin, in-situ carcinoma of the cervix uteri, non-melanomatous skin cancer, carcinoma in situ of the breast, incidental finding of prostate cancer (TNM stage of T1a or T1b), or synchronous H&N primaries
* Currently receiving any other investigational agents.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, nab-paclitaxel, or other agents used in the study. Previous grade 1 or 2 allergic reaction to cetuximab is permissible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 72 hours of start of study treatment.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with the study drugs. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) - with first line therapy | 8 months (estimated median length of treatment)
  PFS is defined as the time from randomization to first radiologic confirmation of disease progression, or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Until death (estimated 24 months)
  OS is defined as the time from randomization to death.
Overall response rate | 8 months (estimated median length of treatment)
  Overall response rate = complete response + partial response
  Evaluated using RECIST 1.1.
Grade 3 and 4 adverse events | 9 months (28 days from last dose of study drug with estimated median length of treatment of 8 months)
  Adverse events will be recorded from the date of first dose of study drug (nab-paclitaxel) until 28 days after the last dose of study drug.
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for all toxicity reporting.
Quality of life | Baseline, End of cycle 2, End of cycle 6, and End of treatment (estimated median length of treatment is 8 months)
  Using the EORTC QLQ-C30, MDADI, FACT-H&N, and FACT/GOG-NTX-4.
  * The EORTC-QLQ-C30 has a total score, one general QOL and one "within the last week" subscale, as well as a single "overall general health" item and a single "overall QOL" item. Scale is from 1-4 with 1 = not at all and 4 = very much on 28 questions. The scale is from 1-7 on 2 questions with 1 = very poor and 7 = excellent.
  * The MDADI has 1 global dysphagia item, physical, function and emotional subscales and one summary scale, which is the sum of the 3 subscales rescaled to 0-100.
  * The FACT instruments have four subscales (physical, social, emotional and functional), as well as 11-12 head and neck cancer-specific questions. The scale goes from 1-4 with 1 = not at all and 4 = very much.
Progression-free survival (PFS) - with maintenance therapy | 8 months (estimated median length of treatment)
  PFS on maintenance therapy is defined as time from first dose of maintenance therapy to first radiologic confirmation of disease progression, or death from any cause.
Disease control | 8 months (estimated median length of treatment)
  Disease control = complete response + partial response + stable disease
  Evaluated using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (5):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Cancer Center Oncology Clinic and Pharmacy, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu